CLINICAL TRIAL: NCT02646449
Title: Treatment of Young Adults With Comorbid AUD/MDD: A Pilot Medication Trial
Acronym: YAAD-P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jack Cornelius, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21AA022863-01A1 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
Keywords: Major Depressive Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Mirtazapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirtazapine (Active Comparator): Gelatin capsules mirtazapine 15 mg, 1 capsule every a.m. Medication will be increased by one capsule, to a dose of 2 capsules barring side effects, at Week 2.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): Gelatin capsules Placebo capsules, identical to mirtazapine capsules, 1 capsule every a.m. Medication will be increased by one capsule to 2 capsules at Week 2, barring any side effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Gelatin capsules mirtazapine 15 mg, 1 capsule every a.m. Medication will be increased by one capsule, to a dose of 2 capsules barring side effects, at Week 2.
  Other Names: Remeron
  Arms: Mirtazapine
Drug: Placebo — Gelatin capsules Placebo capsules, identical to mirtazapine capsules, 1 capsule every a.m. Medication will be increased by one capsule to 2 capsules at Week 2, barring any side effects.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Recent reports have shown that alcohol misuse is a particularly serious problem among the 18 to 25 year old age group. Previous medication trials with SSRI antidepressants among young adults with co-occurring depressive disorders, including our own recent trials with SSRI medications, have produced disappointing results, especially for decreasing the level of alcohol consumption. Mirtazapine is a non-SSRI medication with a unique structure and mechanism of action. Recent study results suggest that mirtazapine is more effective than other antidepressants for treating non-comorbid depression. A few recent studies with mirtazapine have been conducted among subjects with comorbid AUD/MDD, and those studies have demonstrated efficacy for mirtazapine for decreasing the depressive symptoms and the alcohol craving of subjects with comorbid AUD/MDD. However, those studies did not measure level of alcohol consumption, so it is unclear whether mirtazapine decreases the level of alcohol use of that comorbid population. The results of our own very recent open label pilot study suggest robust within-group efficacy for mirtazapine for decreasing both the level of alcohol use and the depressive symptoms of comorbid subjects. However, that pilot study did not include a placebo control group, so the efficacy of mirtazapine versus placebo for decreasing the level of alcohol use among persons with comorbid AUD/MDD remains unclear. This grant submission proposes to conduct a first double-blind, placebo-controlled pilot study to provide a preliminary assessment of the efficacy of mirtazapine versus placebo for decreasing both the alcohol use and depressive symptoms of young adults with comorbid AUD/MDD. If results (effect sizes) from the proposed study are found to be promising concerning outcome differences between the mirtazapine and placebo groups, then we will use those findings to apply for an R01 study to definitively assess the efficacy of mirtazapine for treating young adults with AUD/MDD.

DETAILED DESCRIPTION:
MDD and AUD are each highly prevalent among young adults, and the comorbidity of those two disorders occurs more often than would be expected by chance alone. The presence of this comorbidity is associated with increased risk for motor vehicle accidents, relapse to alcohol use, suicide, recurrence of depressive illness, increased morbidity, and costly hospitalization. Thus, the comorbidity of AUD/MDD is a highly significant public health problem among young adults, with considerable unmet treatment needs. Previous medication trials with SSRI antidepressants involving those co-occurring conditions, including our own recent trials with SSRI medications, have produced disappointing results, especially for decreasing the level of alcohol consumption. Mirtazapine is an FDA-approved medication for treating MDD with a unique pharmacological profile, unrelated to SSRIs. Recent study results suggest that mirtazapine is more effective than other antidepressants for treating non-comorbid depression. A few recent studies have demonstrated efficacy for mirtazapine for decreasing the depressive symptoms and the alcohol craving of subjects with comorbid AUD/MDD, but those studies did not measure level of alcohol consumption. Therefore, it is unclear whether mirtazapine decreases the level of alcohol use of that comorbid population. Our own recent pilot data suggest within-group efficacy for mirtazapine for decreasing both the excessive alcohol use and the depressive symptoms of persons with comorbid AD/MDD. However, that pilot study did not include a placebo control group, so the efficacy of mirtazapine for decreasing the level of alcohol use among persons with comorbid AUD/MDD remains unclear. To date, no double-blind, placebo-controlled study has even been conducted to assess whether mirtazapine decreases both the level of drinking and the depressive symptoms of young adults with comorbid AD/MDD. In this submission, we propose a proof of concept, double-blind, placebo-controlled pilot trial to provide a preliminary assessment of the efficacy of the medication mirtazapine vs. placebo in the treatment of young adults with co-occurring alcohol use disorders (AUD) and major depression (MDD). If results (effect sizes) from the proposed study are found to be promising concerning outcome differences between the mirtazapine and placebo groups, then we will use those findings to apply for an R01 study to definitively assess the efficacy of mirtazapine for treating young adults with AUD/MDD.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR diagnosis of current alcohol dependence, confirmed by the Mini International Neuropsychiatric Interview (MINI)
* DSM-IV-TR diagnosis of current major depressive disorder, confirmed by the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Any person who meets criteria for alcohol-induced depression
* Any psychotic disorder bipolar disorder, mental retardation, impaired cognitive functioning, or use of any psychotropic medication in the previous month
* Current Diagnostic and Statistical Manual (DSM-IV) criteria for dependence on substances other than alcohol, cannabis, nicotine, or caffeine
* Significant neurological conditions or medical conditions
* Persistent elevation of liver function enzymes indicating active liver disease (elevated t. bilirubin or elevation to three-time normal range of liver enzymes, SGOT, SGPT, or g-GTP)
* The presence of renal function impairment defined as serum creatinine >2x upper limit of normal
* Pregnancy, inability or unwillingness to use contraceptive methods
* Use of any antidepressant medication in the prior two months, or any lifetime use of mirtazapine
* Inability to read or understand study forms and agree to informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack R Cornelius, M.D., M.P.H., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornelius JR, Chung T, Douaihy AB, Kirisci L, Glance J, Kmiec J, FitzGerald D, Wesesky MA, Salloum I. Mirtazapine in comorbid major depression and an alcohol use disorder: A double-blind placebo-controlled pilot trial. Psychiatry Res. 2016 Aug 30;242:326-330. doi: 10.1016/j.psychres.2016.06.005. Epub 2016 Jun 15. PMID 27327217

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 11 signed Consent, 7 were started on protocol medications. One patient was excluded after signing consent due to an exclusionary diagnosis (schizophrenia), one due to being over the maximum age limit (patient falsified age at screen), one due to an exclusionary medical diagnosis and one was excluded due to alcohol use under the minimum.
Period: Overall Study
Arm/Group | Mirtazapine | Placebo
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirtazapine | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (1.5) | 24.4 (3.7) | 22.9 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: Level of drinking, as indicated by the number of drinks per day as recorded on the Timeline Follow-Back calendar.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Drinks per drinking day
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 4 | 3
Drinks per drinking day | 2.8 (2.9) | 2.0 (2.0)

2. Primary Outcome: Level of Depressive Symptoms
Description: Level of depressive symptoms, as indicated by the score on the Beck Depression Inventory. The Beck Depression Inventory II scoring range is as follows: 0-13 minimal depressive symptoms, 14-19 mild depressive symptoms, 20-28 moderate depressive symptoms and 29-63 severe depressive symptoms.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirtazapine | Placebo
Number analyzed (Participants) | 4 | 3
units on a scale | 8.0 (14.7) | 3.3 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Baseline Visit through Week 12.
Arm/Group | Mirtazapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No